CLINICAL TRIAL: NCT01259609
Title: Changes in Ciliary Body Thickness in Patients With Diabetic Macular Edema After Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Hyeong Gon Yu, Department of Ophthalmology, Seoul National University Hospital, Seoul, Korea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH_OT
Record Dates: First submitted 2010-12-06; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Ciliary Body; Ultrasound Biomicroscopy; Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diabetic Macular Edema Group (Experimental)
  Interventions: Procedure: Pars Plana Vitrectomy
- Epiretinal Membrane Group (Active Comparator)
  Interventions: Procedure: Pars Plana Vitrectomy
- Healthy Control (No Intervention)

INTERVENTIONS:
Procedure: Pars Plana Vitrectomy — 25-gauge three-port pars plana vitrectomy
  Arms: Diabetic Macular Edema Group; Epiretinal Membrane Group

SUMMARY:
The purpose of this study is to determine whether ciliary body thickness increased in the presence of diabetic macular edema and whether it changed after pars plana vitrectomy.

DETAILED DESCRIPTION:
A diabetic macular edema group consisted of diabetic patients who underwent PPV for diffuse diabetic macular edema. A epiretinal membrane group, a surgical control group, consisted of non-diabetic patients with epiretinal membrane who underwent pars plana vitrectomy. A healthy control was also included for the comparison of preoperative ciliary body thickness. Ciliary body thickness was measured using ultrasound biomicroscopy, and central macular thickness was determined using optical coherence tomography. The visual outcome, ciliary body thickness, and central macular thickness were compared between groups before and 1, 2, and 4 months after pars plana vitrectomy and the correlations between the central macular thickness and ciliary body thickness and best corrected visual acuity were determined.

ELIGIBILITY:
Inclusion Criteria for diabetic macular edema group:

* Diabetic macular edema with preoperative central macular thickness > 300 μm on optical coherence tomography
* Macular edema that was not associated with an epiretinal membrane or traction membrane
* No combined traction retinal detachment or vitreous hemorrhage
* No signs of ocular inflammatory disease on preoperative examination
* Phakic eye
* An axial length between 22.0 mm and 25.0 mm

Exclusion Criteria for diabetic macular edema group:

* Patients with uveitis, inflammatory connective tissue disorders or a history of previous ocular surgery
* Long-term application of topical medication, a history of intravitreal steroid or anti-VEGF injection within 3 months before vitrectomy

Inclusion Criteria for epiretinal membrane group:

* Non-diabetic patients with an epiretinal membrane who were scheduled for vitrectomy
* No ocular or systemic disease other than epiretinal membrane

Inclusion Criteria for healthy group:

* No diabetes
* No ocular disease other than cataract

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
ciliary body thickness | up to four months after surgery
  ciliary body thickness was determined using ultrasound biomicroscopy

SECONDARY OUTCOMES:
central macular thickness | up to four months after surgery
  central macular thickness was determined using optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong Gon Yu, M.D., Principal Investigator — Department of Ophthalmology, Seoul National University Hospital, Seoul, Republic of Korea
Locations (1):
- Department of Ophthalmology, Seoul National University Hospital, Seoul, South Korea